CLINICAL TRIAL: NCT02375464
Title: Gallium-68 DOTATOC for Management of Neuroendocrine Tumors
Status: No longer available | Type: Expanded Access
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Stephen Scharf, Principal Investigator, Northwell Health
Other Study IDs: 15-0587
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine tumor; carcinoid tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor | interventions — Ga(III)-DOTATOC; Gallium-68

INTERVENTIONS:
Drug: Gallium-68 DOTATOC — Imaging with Gallium-68 DOTATOC
  Other Names: Gallium-68 (DOTA0-Phe1-Tyr3)octreotide

SUMMARY:
Gallium-68 DOTATOC is a material used to find neuroendocrine tumors (NETs) using positron emission tomography (PET scan). The material has already been shown to be better than the currently available imaging agents. This study is designed to evaluate the clinical impact of PET CT scanning using this agent in the evaluation and management of patients with NETs.

DETAILED DESCRIPTION:
Patients with NETs will be evaluated by their own physicians. Before doing the PET scan using Gallium-68 DOTATOC, the physicians will be asked to describe the type of treatment that they would recommend. After the test is performed and the result reviewed, the physician will be asked to reevaluate the therapeutic and management options. Data will be analyzed to determine the impact of the testing on patient management.

Gallium-68 has been designated an "orphan drug" due to the relative rarity of NETs. It is expected that the data collected from this and other similar trials will be used to provide data to the FDA regarding the safety and efficacy of this drug as an imaging agent for NETs and ultimately lead to FDA approval.

ELIGIBILITY:
Inclusion Criteria:

* Proven or suspected neuroendocrine tumor Physician referral for imaging

Exclusion Criteria:

* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: STEPHEN C SCHARF, MD, Principal Investigator — Lenox Hill Hospital